CLINICAL TRIAL: NCT06134986
Title: Intermittent Fasting in Adults With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Krista Varady, Professor of Nutrition, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-0678
Record Dates: First submitted 2023-11-11; First posted 2023-11-18 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Time restricted eating (TRE) (Experimental): 8-h eating window Ad libitum food intake from 12-8 pm every day Fasting from 8-12 pm every day (16-h fast)
  Interventions: Other: Time restricted eating
- Daily calorie restriction (CR) (Experimental): 25% energy restriction every day Diet counseling provided
  Interventions: Other: Daily calorie restriction
- Control (No Intervention): Ad libitum food intake, eating over more than 10 hours per day

INTERVENTIONS:
Other: Time restricted eating — 8-h eating window Ad libitum food intake from 12-8 pm every day Fasting from 8-12 pm every day (16-h fast)
  Arms: Time restricted eating (TRE)
Other: Daily calorie restriction — 25% energy restriction every day Diet counseling provided
  Arms: Daily calorie restriction (CR)

SUMMARY:
The majority of adults with type 1 diabetes (T1DM) have either overweight or obesity. As such, dietary management has been recommended as an adjunct to insulin treatment to improve glycemic control and facilitate weight loss in patients with T1DM. Daily calorie restriction (CR) is the main diet prescribed to patients with T1DM for weight loss. However, many patients find it difficult to adhere to CR because calorie intake must be vigilantly monitored every day. In light of these problems with CR, another approach that limits timing of food intake, instead of number of calories consumed, has been developed. This diet is called "time restricted eating" (TRE) and involves confining the period of food intake to 6-8 h per day. TRE allows individuals to self-select foods and eat ad libitum during a large part of the day, which greatly increases compliance to these protocols. The simplicity of TRE, its accommodation of dietary preferences, and associated weight loss may translate to improved glycemic measures in patients with T1DM. The present study will be the first randomized controlled trial to compare the effect of TRE versus CR for weight management and improved glycemic control in adults with obesity and T1DM.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 75 years old
* BMI between 25 and 50 kg/m2
* Previously diagnosed with T1DM and currently using insulin
* HbA1c: 6.5-9.5% (regardless of medication use)
* On either multiple daily doses of insulin (MDI) program or using an insulin pump (with or without closed loop feature) 11
* Active prescription for glucagon

Exclusion Criteria:

* Previously diagnosed with T2DM
* Have a history of eating disorders (anorexia, bulimia, or binge eating disorder)
* Are not weight stable for 3 months prior to the beginning of study (weight gain or loss > 4 kg)
* Are not able to keep a food diary for 7 consecutive days during screening
* Are eating less than a 10-hour window at baseline
* Are pregnant, or trying to become pregnant
* Are night shift workers
* History of severe hypoglycemia defined as requiring help from others, needed to use emergency glucagon administration in the past 6 months.
* Other significant medical history including heart failure, unstable coronary artery disease, chronic obstructive pulmonary disease requiring oxygen, cirrhosis, active cancer, history of stroke, end stage renal disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Change in percent body weight | Measured at baseline and month 6
  Measured by an electronic scale

SECONDARY OUTCOMES:
Change in HbA1c | Measured at baseline and month 6
  Measured by outside lab (Medstar, IN)
Change in total time in euglycemic range | Measured at baseline and month 6
  Measured by continuous glucose monitor (CGM)
Change in mean glucose level | Measured at baseline and month 6
  Measured by continuous glucose monitor (CGM)
Change in standard deviation of glucose level | Measured at baseline and month 6
  Measured by continuous glucose monitor (CGM)
Change in coefficient of variation of glucose level | Measured at baseline and month 6
  Measured by continuous glucose monitor (CGM)
Change fasting glucose | Measured at baseline and month 6
  Measured by outside lab (Medstar, IN)
Change in absolute body weight | Measured at baseline and month 6
  Measured by an electronic scale
Change in fat mass, lean mass, visceral fat mass | Measured at baseline and month 6
  Measured by DXA
Change in waist circumference | Measured at baseline and month 6
  Measured by measuring tape
Change in body mass index (BMI) | Measured at baseline and month 6
  Calculated as kg/meter squared
Change in plasma lipids (total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides) | Measured at baseline and month 6
  Measured by outside lab (Medstar, IN)
Change in systolic and diastolic blood pressure | Measured at baseline and month 6
  Measured by blood pressure cuff
Change in heart rate | Measured at baseline and month 6
  Measured by blood pressure cuff
Change in energy and nutrient intake | Measured at baseline and month 6
  Measured by 7-day food record
Change in dietary adherence | Measured at baseline and month 6
  Measured by 7-day food record and adherence log
Change in physical activity (steps/d) | Measured at baseline and month 6
  Measured by activity monitor
Adverse events | Measured at baseline and month 6
  Measured by adverse events survey
Change in medication effect score (MES) | Measured at baseline and month 6
  Measured by survey. Total score 0-100. Lower scores indicate less medication used, higher scores indicate more medication used.
Change in ketones | Measured at baseline and month 6
  Measured by ketone meter

CONTACTS AND LOCATIONS:
Overall Officials: Krista Varady, PhD, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No